CLINICAL TRIAL: NCT01442324
Title: Studio Clinico Pilota Con Uso di Elettroporazione Irreversibile (IRE) Nel Trattamento di Lesioni Neoplastiche Epatiche Con Localizzazione ad accessibilità Limitata o ad Alto Rischio
Brief Title: Pilot Study of Irreversible Electroporation (IRE) to Treat Metastatic Liver Cancer & Cholangiocarcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Azienda Ospedaliera di Padova (Other)
Responsible Party: Principal Investigator, Prof. Umberto Cillo, Director of the Hepatobiliary Surgery and Liver Transplantation Unit, Azienda Ospedaliera di Padova
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2252P
Record Dates: First submitted 2011-09-27; First posted 2011-09-28 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Metastatic Liver Cancer; Cholangiocarcinoma; Neoplasm Metastasis
Keywords: Laparotomic surgery; Laparoscopic surgery; Percutaneos tumour ablation; Irreversible electroporation (IRE)
MeSH Terms: conditions — Liver Neoplasms; Cholangiocarcinoma; Neoplasm Metastasis | interventions — Electroporation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IRE (Experimental): Patients will be subjected to irreversible electroporation (IRE) as the sole treatment of nodules not considered treatable by resection or thermal ablation.
  Interventions: Procedure: Irreversible electroporation (IRE)

INTERVENTIONS:
Procedure: Irreversible electroporation (IRE) — Needle-like electrodes are inserted through the liver and in the lesion without exceeding its deepest margin, at which point the IRE NanoKnife™ System (AngioDynamics) is started.
  Other Names: NanoKnife™ System; AngioDynamics

SUMMARY:
Single-arm pilot clinical trial. Patients will be subjected to irreversible electroporation (IRE) as the sole treatment of nodules not considered treatable by resection or thermal ablation.

DETAILED DESCRIPTION:
Single-arm pilot clinical trial. Patients will be subjected to irreversible electroporation (IRE) as the sole treatment of nodules not considered treatable by resection or thermal ablation.

This pilot study was designed to study the feasibility and safety of treatment as an alternative therapeutic IRE in the treatment of neoplastic nodules in the liver, with particular reference to metastatic liver cancer and cholangiocarcinoma, where the current therapeutic arsenal is inadequate or counter-indicated.

To perform the IRE procedure the IRE NanoKnife™ System (AngioDynamics) will be used.

ELIGIBILITY:
Inclusion Criteria:

* older than 18 years,
* male or female,
* diagnosis of secondary liver cancer or cholangiocarcinoma based on positive biopsy or noninvasive criteria,
* presence of at least one lesion untreatable by surgical resection or ablation for microwave or radio frequency,
* the target nodule must have a diameter of ≤ 5 cm
* ECOG score(Eastern Cooperative Oncology Group) 0,
* ASA score (American Society of Anesthesiologists) ≤ 3,
* prothrombin time ratio >50%
* platelet count >50x10^9/l,
* patient's ability to discontinue anticoagulant and antiplatelet therapy for seven days before and seven days after surgery with NanoKnife™,
* ability to understand and willingness to sign the written informed consent form (ICF),
* life expectancy of at least 3 months.

Exclusion Criteria:

* presence of more than 5 liver lesions,
* previous treatment of the target nodule,
* patient received systemic chemotherapy within 30 days of treatment with the IRE NanoKnife™,
* heart failure, coronary artery disease or arrhythmia in progress, active implantable devices (eg pacemaker),
* pregnant women or women of childbearing potential not using an acceptable method of contraception,
* patient undergoing treatment with an investigational drug within 30 days of treatment with the IRE NanoKnife™,
* in the opinion of the researcher, anyone who can not follow the calendar of visits and assessments of the Protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of IRE for the treatment of metastatic liver cancer or cholangiocarcinoma. | 1 month post-intervention
  The primary measurement parameter for the purposes of this determination is the evaluation of the response of IRE treated lesions according to modified RECIST criteria using CT images or magnetic resonance imaging performed 20 to 40 days after treatment.

SECONDARY OUTCOMES:
Safety | 30 days post-intervention
  The safety endpoint will be the occurrence of serious adverse events related to treatment within 30 days of treatment. All adverse events will be classified according to CTCAE version 3.0 criteria.
Time to in situ recurrence | 2 years post-intervention

CONTACTS AND LOCATIONS:
Overall Officials: Umberto Cillo, MD, Study Chair — Azienda Ospedaliera di Padova; Alessandro Vitale, MD, Principal Investigator — Azienda Ospedaliera di Padova
Locations (1):
- Azienda Ospedaliera di Padova, Padua, PD, Italy

REFERENCES:
- [Background] Ball C, Thomson KR, Kavnoudias H. Irreversible electroporation: a new challenge in "out of operating theater" anesthesia. Anesth Analg. 2010 May 1;110(5):1305-9. doi: 10.1213/ANE.0b013e3181d27b30. Epub 2010 Feb 8. PMID 20142349
- [Background] Onik G, Mikus P, Rubinsky B. Irreversible electroporation: implications for prostate ablation. Technol Cancer Res Treat. 2007 Aug;6(4):295-300. doi: 10.1177/153303460700600405. PMID 17668936
- [Background] Esser AT, Smith KC, Gowrishankar TR, Weaver JC. Towards solid tumor treatment by irreversible electroporation: intrinsic redistribution of fields and currents in tissue. Technol Cancer Res Treat. 2007 Aug;6(4):261-74. doi: 10.1177/153303460700600402. PMID 17668933
- [Background] Al-Sakere B, Andre F, Bernat C, Connault E, Opolon P, Davalos RV, Rubinsky B, Mir LM. Tumor ablation with irreversible electroporation. PLoS One. 2007 Nov 7;2(11):e1135. doi: 10.1371/journal.pone.0001135. PMID 17989772
- See also: Hepatobiliary surgery and Liver Transplantation Unit, University Hospital of Padua (Italy) — http://www.fegatochirurgia.com